CLINICAL TRIAL: NCT01632345
Title: Multicenter, Double-Blind, Randomized, 2-Part, Dose Ranging Study to Compare the Safety, and Antiretroviral Activity of MK-1439 Plus TRUVADA Versus Efavirenz Plus TRUVADA in Antiretroviral Treatment-Naive, HIV-1 Infected Patients
Brief Title: A Dose-Ranging Study to Compare Doravirine (MK-1439) Plus TRUVADA® Versus Efavirenz Plus TRUVADA® in Human Immunodeficiency Virus (HIV)-1 Infected Participants (MK-1439-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1439-007; MK-1439-007 (Other: Merck); 2012-001573-93 (EudraCT Number)
Record Dates: First submitted 2012-06-28; First posted 2012-07-02 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — doravirine; efavirenz; Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Doravirine 25 mg (Experimental): Doravirine 25 mg + TRUVADA® Participants in this arm will receive doravirine 25 mg in Part I and the selected doravirine dose (either 25 mg, 50 mg, 100 mg, or 200 mg) in Part II. These participants also receive placebo that matches efavirenz.
  Interventions: Drug: Doravirine; Drug: TRUVADA®; Drug: Placebo for Doravirine
- Doravirine 50 mg (Experimental): Doravirine 50 mg + TRUVADA® Participants in this arm will receive doravirine 50 mg in Part I and the selected doravirine dose (either 25 mg, 50 mg, 100 mg, or 200 mg) in Part II. These participants also receive placebo that matches efavirenz.
  Interventions: Drug: Doravirine; Drug: TRUVADA®; Drug: Placebo for Doravirine
- Doravirine 100 mg (Experimental): Doravirine 100 mg + TRUVADA® Participants in this arm will receive doravirine 100 mg in Part I and the selected doravirine dose (either 25 mg, 50 mg, 100 mg, or 200 mg) in Part II. These participants also receive placebo that matches efavirenz.
  Interventions: Drug: Doravirine; Drug: TRUVADA®; Drug: Placebo for Doravirine
- Doravirine 200 mg (Experimental): Doravirine 200 mg + TRUVADA® Participants in this arm will receive doravirine 200 mg in Part I and the selected doravirine dose (either 25 mg, 50 mg, 100 mg, or 200 mg) in Part II. These participants also receive placebo that matches efavirenz.
  Interventions: Drug: Doravirine; Drug: TRUVADA®; Drug: Placebo for Doravirine
- Efavirenz (Active Comparator): Efavirenz + TRUVADA® Participants in this arm will receive efavirenz in Part I and in Part II. These participants also receive placebo that matches doravirine.
  Interventions: Drug: Efavirenz; Drug: TRUVADA®; Drug: Placebo for Efavirenz

INTERVENTIONS:
Drug: Doravirine — Part I: Doravirine 25 mg, 50 mg (25 mg X 2), 100 mg, or 200 mg (100 mg X 2) depending upon randomization, taken orally every morning with or without food for at least 24 weeks. Part II: Selected dose of doravirine depending upon randomization (either 25 mg, 50 mg, 100 mg, or 200 mg) tablet orally every morning with or without food for 96 weeks.
  Other Names: MK-1439
  Arms: Doravirine 100 mg; Doravirine 200 mg; Doravirine 25 mg; Doravirine 50 mg
Drug: Efavirenz — Efavirenz 600 mg tablet orally at bedtime taken without food on an empty stomach for 96 weeks
  Arms: Efavirenz
Drug: TRUVADA® — Open-label TRUVADA® (fixed combination 200 mg emtricitabine and 300 mg tenofovir disoproxil fumarate) tablet taken orally with food in the morning for 96 weeks
Drug: Placebo for Doravirine — Placebo tablets matching doravirine
  Arms: Doravirine 100 mg; Doravirine 200 mg; Doravirine 25 mg; Doravirine 50 mg
Drug: Placebo for Efavirenz — Placebo tablets matching efavirenz
  Arms: Efavirenz

SUMMARY:
The hypothesis tested in this study is that doravirine (MK-1439) at the final dose selected is superior to efavirenz, each given in combination with TRUVADA®, as measured by the percentage of participants with CNS events by Week 8. If superiority is established at Week 8, the same hypothesis will be tested for Week 24.

DETAILED DESCRIPTION:
Part I - Dose-Ranging. Part I will evaluate the (1) safety and tolerability and (2) efficacy (antiretroviral activity) of 4 doses of doravirine compared with efavirenz, when each is given in combination with TRUVADA® for at least 24 weeks in approximately 200 participants. A single dose of doravirine will be selected for further study after all participants complete the Week 24 visit in Part I. Participants receiving any dose of doravirine in Part I will be switched to the selected doravirine dose and continue in the study for up to 96 weeks, but will not be randomized to Part II.

Part II - Selected Dose. Part II will be initiated after the doravirine dose has been selected as indicated above for Part 1. Approximately 120 additional participants will be randomized in 1:1 ratio to the selected dose of doravirine or efavirenz, each in combination with TRUVADA® for 96 weeks of blinded treatment. Part II will evaluate the safety of the selected dose compared with efavirenz, particularly with regard to central nervous system (CNS) adverse events.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive
* No previous use of antiretroviral therapy (ART)
* No signs of active pulmonary disease within 45 days before the start of study treatment
* Clinically stable with no signs or symptoms of acute infection
* No change in clinical status or chronic medications for at least 2 weeks before the start of study treatment
* Participants of reproductive potential agree to remain abstinent in line with their preferred and usual lifestyle or use (or have their partner use) 2 acceptable methods of birth control throughout the study and for 12 weeks post study.
* Participants not of reproductive potential, not sexually active, whose current partner(s) is not of reproductive potential, or whose sexual activity is exclusively homosexual are eligible without requiring the use of contraception.

Exclusion Criteria:

* Males planning to impregnate or provide sperm donation for the duration of the study plus an additional 12 weeks. Females pregnant or breast-feeding or expecting to conceive or donate eggs for the duration of the study plus an additional 12 weeks.
* Received any approved or experimental antiretroviral agents or is anticipated to receive such medications during the study.
* Use of any immunomodulators or immunosuppressive therapy within one month before the study. Short courses of corticosteroids (e.g., for asthma exacerbation) are allowed.
* Treatment for a viral infection other than HIV, such as hepatitis B, with an agent that is active against HIV
* HIV resistance to emtricitabine, tenofovir disoproxil fumarate, and/or efavirenz.
* History of renal or urinary obstructive disease or requires dialysis
* Active Hepatitis C virus (HCV) or Hepatitis B virus (HBV) co-infection
* History of alcohol or other substance abuse
* Participation in a study with an investigational compound/device within one month or is anticipating to participate in such a study during this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2012-10-12 (Actual); Primary Completion 2014-12-03 (Actual); Study Completion 2016-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Gatell JM, Morales-Ramirez JO, Hagins DP, Thompson M, Arasteh K, Hoffmann C, Raffi F, Osiyemi O, Dretler R, Harvey C, Xu X, Plettenberg A, Smith DE, Portilla J, Rugina S, Kumar S, Frobose C, Wan H, Rodgers A, Hwang C, Teppler H. Doravirine dose selection and 96-week safety and efficacy versus efavirenz in antiretroviral therapy-naive adults with HIV-1 infection in a Phase IIb trial. Antivir Ther. 2019;24(6):425-435. doi: 10.3851/IMP3323. PMID 31355775
- [Derived] Thompson M, Orkin C, Molina JM, Sax P, Cahn P, Squires K, Xu X, Rodgers A, Kumar S, Teppler H, Martin E, Hanna G, Hwang C. Once-daily Doravirine for Initial Treatment of Adults Living With Human Immunodeficiency Virus-1: An Integrated Safety Analysis. Clin Infect Dis. 2020 Mar 17;70(7):1336-1343. doi: 10.1093/cid/ciz423. PMID 31121013

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 210 participants were randomized to Part I and 132 participants were randomized to Part II.
Groups:
- Part I: Doravirine 25 mg: Doravirine 25 mg once daily plus TRUVADA once daily in Part I
- Part I: Doravirine 50 mg: Doravirine 50 mg once daily plus TRUVADA once daily in Part I
- Part I: Doravirine 100 mg: Doravirine 100 mg once daily plus TRUVADA once daily in Part I
- Part I: Doravirine 200 mg: Doravirine 200 mg once daily plus TRUVADA once daily in Part I
- Part I: Efavirenz 600 mg: Efavirenz 600 mg once daily plus TRUVADA once daily in Part I
- Part II: Doravirine 100 mg: Doravirine 100 mg once daily plus TRUVADA once daily in Part II
- Part II: Efavirenz 600 mg: Efavirenz 600 mg once daily plus TRUVADA once daily in Part II
Period: Randomized Participants
Arm/Group | Part I: Doravirine 25 mg | Part I: Doravirine 50 mg | Part I: Doravirine 100 mg | Part I: Doravirine 200 mg | Part I: Efavirenz 600 mg | Part II: Doravirine 100 mg | Part II: Efavirenz 600 mg
Started | 41 | 43 | 42 | 41 | 43 | 66 | 66
Completed | 41 | 43 | 42 | 41 | 43 | 66 | 66
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment: Part I
Arm/Group | Part I: Doravirine 25 mg | Part I: Doravirine 50 mg | Part I: Doravirine 100 mg | Part I: Doravirine 200 mg | Part I: Efavirenz 600 mg | Part II: Doravirine 100 mg | Part II: Efavirenz 600 mg
Started | 41 | 43 | 42 | 41 | 43 | 0 (Participants in Part II did not participate in Part I.) | 0 (Participants in Part II did not participate in Part I.)
Treated | 40 | 43 | 42 | 41 | 43 | 0 | 0
Completed | 29 | 28 | 32 | 33 | 30 | 0 | 0
Not Completed | 12 | 15 | 10 | 8 | 13 | 0 | 0
Not completed — Adverse Event | 1 | 4 | 2 | 1 | 3 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 3 | 2 | 1 | 3 | 4 | 0 | 0
Not completed — Non-Compliance with Study Drug | 3 | 2 | 2 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 2 | 1 | 0 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 4 | 4 | 1 | 4 | 0 | 0
Period: Treatment: Part II
Arm/Group | Part I: Doravirine 25 mg | Part I: Doravirine 50 mg | Part I: Doravirine 100 mg | Part I: Doravirine 200 mg | Part I: Efavirenz 600 mg | Part II: Doravirine 100 mg | Part II: Efavirenz 600 mg
Started | 0 (Participants in Part I did not continue in Part II.) | 0 (Participants in Part I did not continue in Part II.) | 0 (Participants in Part I did not continue in Part II.) | 0 (Participants in Part I did not continue in Part II.) | 0 (Participants in Part I did not continue in Part II.) | 66 (66 new participants enrolled at 100 mg dose in Part II.) | 66 (66 new participants enrolled at efavirenz treatment in Part II.)
Treated | 0 | 0 | 0 | 0 | 0 | 66 | 66
Completed | 0 | 0 | 0 | 0 | 0 | 55 | 55
Not Completed | 0 | 0 | 0 | 0 | 0 | 11 | 11
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 3 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 3 | 1
Not completed — Non-Compliance with Study Drug | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Population: All Treated participants randomized to doravirine or efavirenz using an interactive voice response system (IVRS)
Groups:
- Doravirine 25 mg: Part I/II Combined: Doravirine 25 mg once daily plus TRUVADA once daily
- Doravirine 50 mg Part I/II Combined: Doravirine 50 mg once daily plus TRUVADA once daily
- Doravirine 100 mg: Part I/II Combined: Doravirine 100 mg once daily plus TRUVADA once daily
- Doravirine 200 mg: Part I/II Combined: Doravirine 200 mg once daily plus TRUVADA once daily
- Efavirenz 600 mg: Part I/II Combined: Efavirenz 600 mg once daily plus TRUVADA once daily
- Total: Total of all reporting groups
Arm/Group | Doravirine 25 mg: Part I/II Combined | Doravirine 50 mg Part I/II Combined | Doravirine 100 mg: Part I/II Combined | Doravirine 200 mg: Part I/II Combined | Efavirenz 600 mg: Part I/II Combined | Total
Number analyzed (Participants) | 40 | 43 | 108 | 41 | 108 | 340
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (13.42) | 38.3 (10.71) | 36.8 (11.31) | 34.4 (8.85) | 35.2 (9.08) | 36.4 (10.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 6 | 9 | 1 | 7 | 25
  Male | 38 | 37 | 99 | 40 | 101 | 315

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least 1 AE in Weeks 0-24: Doravirine (All Doses) vs Efavirenz (Part I)
Description: Assessment of the percentage of participants receiving doravirine at all doses (25 mg, 50 mg, 100 mg, or 200 mg), compared with participants receiving efavirenz 600 mg, who had at least 1 AE over 24 weeks of treatment. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product.The percentage of participants in any treatment group with at least 1 AE was primarily assessed for Weeks 0-24.
Time Frame: Up to Week 24
Population: The analyzed population consisted of all randomized participants who received at least 1 dose of study treatment in Part I.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Doravirine 25 mg: Part I: Doravirine 25 mg once daily plus TRUVADA once daily received in Part I
- Doravirine 50 mg: Part I: Doravirine 50 mg once daily plus TRUVADA once daily received in Part I
- Doravirine 100 mg : Part I: Doravirine 100 mg once daily plus TRUVADA once daily received in Part I
- Doravirine 200 mg: Part I: Doravirine 200 mg once daily plus TRUVADA once daily received in Part I
- Efavirenz 600 mg: Part I: Efavirenz 600 mg once daily plus TRUVADA once daily received in Part I
Arm/Group | Doravirine 25 mg: Part I | Doravirine 50 mg: Part I | Doravirine 100 mg : Part I | Doravirine 200 mg: Part I | Efavirenz 600 mg: Part I
Number analyzed (Participants) | 40 | 43 | 42 | 41 | 42
Percentage of participants | 90.0 [76.3 to 97.2] | 93.0 [80.9 to 98.5] | 71.4 [55.4 to 84.3] | 85.4 [70.8 to 94.4] | 83.3 [68.6 to 93.0]
Statistical Analysis 1: Comparison: Doravirine 25 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference (Doravirine - Efavirenz) = 6.7, 95% CI 2-sided [-9.0 to 22.4] — A negative value would be considered as favoring doravirine over efavirenz
Statistical Analysis 2: Comparison: Doravirine 50 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference (Doravirine - Efavirenz) = 9.7, 95% CI 2-sided [-4.6 to 24.9] — A negative value would be considered as favoring doravirine over efavirenz
Statistical Analysis 3: Comparison: Doravirine 100 mg : Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference (Doravirine - Efavirenz) = -11.9, 95% CI 2-sided [-27.9 to 6.3] — A negative value would be considered as favoring doravirine over efavirenz
Statistical Analysis 4: Comparison: Doravirine 200 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference (Doravirine - Efavirenz) = 2.0, 95% CI 2-sided [-14.5 to 18.4] — A negative value would be considered as favoring doravirine over efavirenz

2. Primary Outcome: Percentage of Participants Who Discontinued Study Therapy Due to AEs in Weeks 0-24: Doravirine (All Doses) vs Efavirenz (Part I)
Description: Assessment of the percentage of participants receiving doravirine at all doses (25 mg, 50 mg, 100 mg, or 200 mg), compared with participants receiving efavirenz 600 mg, who discontinued therapy due to an AE over 24 weeks of treatment. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product.The percentage of participants in any treatment group who discontinued therapy due to an AE was primarily assessed for Weeks 0-24.
Time Frame: Up to Week 24
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Doravirine 100 mg: Part I: Doravirine 100 mg once daily plus TRUVADA once daily received in Part I
Arm/Group | Doravirine 25 mg: Part I | Doravirine 50 mg: Part I | Doravirine 100 mg: Part I | Doravirine 200 mg: Part I | Efavirenz 600 mg: Part I
Number analyzed (Participants) | 40 | 43 | 42 | 41 | 42
Percentage of participants | 2.5 [0.1 to 13.2] | 7.0 [1.5 to 19.1] | 2.4 [0.1 to 12.6] | 0.0 [0.0 to 8.6] | 4.8 [0.6 to 16.2]
Statistical Analysis 1: Comparison: Doravirine 25 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference (Doravirine - Efavirenz) = -2.3, 95% CI 2-sided [-13.7 to 8.8] — A negative value would be considered as favoring doravirine over efavirenz
Statistical Analysis 2: Comparison: Doravirine 50 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference (Doravirine - Efavirenz) = 2.2, 95% CI 2-sided [-9.9 to 14.7] — A negative value would be considered as favoring doravirine over efavirenz
Statistical Analysis 3: Comparison: Doravirine 100 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference (Doravirine - Efavirenz) = -2.4, 95% CI 2-sided [-13.8 to 8.2] — A negative value would be considered as favoring doravirine over efavirenz
Statistical Analysis 4: Comparison: Doravirine 200 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference (Doravirine - Efavirenz) = -4.8, 95% CI 2-sided [-15.9 to 4.1] — A negative value would be considered as favoring doravirine over efavirenz

3. Primary Outcome: Percentage of Participants With At Least 1 AE in Weeks 0-24: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: Assessment of the percentage of participants receiving doravirine at 100 mg, compared with participants receiving efavirenz 600 mg, who had at least 1 AE over 24 weeks of treatment. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product.The percentage of participants in any treatment group with at least 1 AE was assessed for Weeks 0-24.
Time Frame: Up to Week 24
Population: The analyzed population consisted of all randomized participants who received at least 1 dose of study treatment in either Part I or Part II.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- Doravirine 100 mg: Part I/II (Combined): Doravirine 100 mg once daily plus TRUVADA once daily received in either Part I or Part II
- Efavirenz 600 mg: Part I/II (Combined): Efavirenz 600 mg once daily plus TRUVADA once daily received in either Part I or Part II
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 108 | 108
Percentage of participants | 75.0 [65.7 to 82.8] | 85.2 [77.1 to 91.3]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference = -10.2, 95% CI 2-sided [-20.9 to 0.5] — A negative value would be considered as favoring doravirine over efavirenz

4. Primary Outcome: Percentage of Participants With CNS Events by Week 8: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: Assessment of the percentage of participants receiving doravirine at 100 mg, compared with participants receiving efavirenz 600 mg, who had CNS events over 8 weeks of treatment. CNS events were pooled and evaluated as pre-specified by the protocol (depression, nightmare, confusional state, suicidal ideation, nervous system disorder, psychotic disorder, abnormal dreams, suicide attempt, acute psychosis, delirium, depressed level of consciousness, hallucination, hallucination auditory, hallucination visual, completed suicide, suicidal behavior, major depression, depressed mood, depressive symptom, insomnia, disturbance in attention, somnolence, dizziness, or concentration impaired). The percentage of participants in either treatment group with CNS events was assessed over Weeks 0-8.
Time Frame: Up to Week 8
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 108 | 108
Percentage of participants | 24.1 [16.4 to 33.3] | 44.4 [34.9 to 54.3]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; p = 0.002, Miettinen and Nurminen method — Superiority analysis; Difference (Doravirine - Efavirenz) = -20.4, 95% CI 2-sided [-32.4 to -7.8] — A negative value would be considered as favoring doravirine over efavirenz

5. Primary Outcome: Percentage of Participants With CNS Events by Week 24: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: Assessment of the percentage of participants receiving doravirine at 100 mg, compared with participants receiving efavirenz 600 mg, who had CNS events over 24 weeks of treatment. CNS events were pooled and evaluated as pre-specified by the protocol (depression, nightmare, confusional state, suicidal ideation, nervous system disorder, psychotic disorder, abnormal dreams, suicide attempt, acute psychosis, delirium, depressed level of consciousness, hallucination, hallucination auditory, hallucination visual, completed suicide, suicidal behavior, major depression, depressed mood, depressive symptom, insomnia, disturbance in attention, somnolence, dizziness, or concentration impaired). The percentage of participants in either treatment group with CNS events was assessed over Weeks 0-24.
Time Frame: Up to Week 24
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 108 | 108
Percentage of participants | 26.9 [18.8 to 36.2] | 47.2 [37.5 to 57.1]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; p = 0.002, Miettinen and Nurminen method — Superiority analysis; Difference (Doravirine - Efavirenz) = -20.4, 95% CI 2-sided [-32.6 to -7.5] — A negative value would be considered as favoring doravirine over efavirenz

6. Primary Outcome: Percentage of Participants With Virologic Response (HIV-1 RNA) < 40 Copies/mL) at Week 24: Doravirine (All Doses) vs Efavirenz (Part I)
Description: Assessment of the virologic response to doravirine at all studied doses (25 mg, 50 mg, 100 mg, and 200 mg), compared to efavirenz, each in combination with TRUVADA, as measured by the percentage of participants with plasma HIV-1 RNA <40 copies/mL at Week 24. HIV RNA levels were determined using the Abbott RealTime HIV-1 Assay, which has a limit of reliable quantification of 40 copies/mL. The percentage of participants in any treatment group with a virologic response was assessed at Week 24. The Non-Completer = Failure (NC=F) approach, in which participants who prematurely discontinued assigned treatment for any reason and were considered as failures thereafter, was used as the primary approach to handle missing data this analysis of efficacy.This primary outcome was analyzed for HIV-1 RNA <40 copies/mL in Part I.
Time Frame: Week 24
Population: The analyzed population consisted of all randomized participants who received at least one dose of blinded study treatment in Part I, and had at least one post-randomization observation for the analysis of HIV-1 RNA (<40 copies/mL) at 24 weeks of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 25 mg: Part I | Doravirine 50 mg: Part I | Doravirine 100 mg: Part I | Doravirine 200 mg: Part I | Efavirenz 600 mg: Part I
Number analyzed (Participants) | 40 | 43 | 42 | 41 | 42
Percentage of participants | 80.0 [64.4 to 90.9] | 74.4 [58.8 to 86.5] | 71.4 [55.4 to 84.3] | 80.5 [65.1 to 91.2] | 64.3 [48.0 to 78.4]
Statistical Analysis 1: Comparison: Doravirine 25 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in % response = 15.7, 95% CI 2-sided [-4.1 to 34.4] — A positive value would be considered as favoring doravirine over efavirenz
Statistical Analysis 2: Comparison: Doravirine 50 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in % response = 10.0, 95% CI 2-sided [-9.6 to 29.1] — A positive value would be considered as favoring doravirine over efavirenz
Statistical Analysis 3: Comparison: Doravirine 100 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in % response = 6.6, 95% CI 2-sided [-13.2 to 26.0] — A positive value would be considered as favoring doravirine over efavirenz
Statistical Analysis 4: Comparison: Doravirine 200 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in % response = 15.9, 95% CI 2-sided [-3.4 to 34.4] — A positive value would be considered as favoring doravirine over efavirenz

7. Primary Outcome: Percentage of Participants With Virologic Response (HIV-1 RNA <40 Copies/mL) at Week 24: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: Assessment of the virologic response to doravirine at 100 mg, compared to efavirenz, each in combination with TRUVADA, as measured by the percentage of participants with HIV-1 RNA <40 copies/mL at Week 24. HIV RNA levels were determined using the Abbott RealTime HIV-1 Assay, which has a limit of reliable quantification of 40 copies/mL. The percentage of participants in any treatment group with a virologic response was assessed at Week 24. The NC=F approach was used as the primary approach to handle missing data this analysis of efficacy. This primary outcome was analyzed for HIV-1 RNA <40 copies/mL in Part I & Part II combined.
Time Frame: Week 24
Population: The analyzed population consisted of all randomized participants who received at least one dose of blinded study treatment in either Part I or Part II, and had at least one post-randomization observation for the analysis of HIV-1 RNA (<40 copies/mL) at 24 weeks of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 107 | 108
Percentage of participants | 72.9 [63.4 to 81.0] | 73.1 [63.8 to 81.2]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference in % response = -0.5, 95% CI 2-sided [-13.2 to 11.2] — A positive value would be considered as favoring doravirine over efavirenz

8. Secondary Outcome: Percentage of Participants With Virologic Response (HIV-1 RNA <40 Copies/mL) at Week 48: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: Assessment of the virologic response to doravirine at 100 mg, compared to efavirenz, each in combination with TRUVADA, as measured by the percentage of participants with HIV-1 RNA <40 copies/mL at Week 48. HIV RNA levels were determined using the Abbott RealTime HIV-1 Assay. The percentage of participants in any treatment group with a virologic response was primarily assessed for Weeks 0-24. The NC=F approach was used as the primary approach to handle missing data this analysis of efficacy. This primary outcome was analyzed for HIV-1 RNA <40 copies/mL in Part I & Part II combined.
Time Frame: Week 48
Population: The analyzed population consisted of all randomized participants who received at least one dose of blinded study treatment in either Part I or Part II, and had at least one post-randomization observation for the analysis of HIV-1 RNA (<40 copies/mL) at 48 weeks of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 77.8 [68.8 to 85.2] | 79.4 [70.5 to 86.6]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference in % response = -1.9, 95% CI 2-sided [-12.9 to 9.2] — A positive value would be considered as favoring doravirine over efavirenz

9. Secondary Outcome: Percentage of Participants With Virologic Response (HIV-1 RNA <40 Copies/mL) at Week 96: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: Assessment of the virologic response to doravirine at 100 mg, compared to efavirenz, each in combination with TRUVADA, as measured by the percentage of participants with HIV-1 RNA <40 copies/mL at Week 96. HIV RNA levels were determined using the Abbott RealTime HIV-1 Assay. The percentage of participants in any treatment group with a virologic response was primarily assessed for Weeks 0-24. The NC=F approach was used as the primary approach to handle missing data this analysis of efficacy. This primary outcome was analyzed for HIV-1 RNA <40 copies/mL in Part I & Part II combined.
Time Frame: Week 96
Population: The analyzed population consisted of all randomized participants who received at least one dose of blinded study treatment in either Part I or Part II, and had at least one post-randomization observation for the analysis of HIV-1 RNA (<40 copies/mL) at 96 weeks of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 108 | 108
Percentage of participants | 75.0 [65.7 to 82.8] | 75.9 [66.7 to 83.6]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference in % response = -0.8, 95% CI 2-sided [-12.4 to 10.7] — A positive value would be considered as favoring doravirine over efavirenz

10. Secondary Outcome: Percentage of Participants With Virologic Response (HIV-1 RNA <200 Copies/mL) at Week 24: Doravirine (All Doses) vs Efavirenz (Part I)
Description: Assessment of the virologic response to doravirine at all studied doses (25 mg, 50 mg, 100 mg, and 200 mg), compared to efavirenz, each in combination with TRUVADA, as measured by the percentage of participants with plasma HIV-1 RNA <200 copies/mL at Week 24. HIV RNA levels were determined using the Abbott RealTime HIV-1 Assay.The percentage of participants in any treatment group with a virologic response was assessed at Week 24. The NC=F approach was used as the primary approach to handle missing data for this analysis of efficacy. This primary outcome was analyzed for HIV-1 RNA <200 copies/mL in Part I.
Time Frame: Week 24
Population: The analyzed population consisted of all randomized participants who received at least one dose of blinded study treatment in Part I, and had at least one post-randomization observation for the analysis of HIV-1 RNA (<200 copies/mL) at 24 weeks of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 25 mg: Part I | Doravirine 50 mg: Part I | Doravirine 100 mg: Part I | Doravirine 200 mg: Part I | Efavirenz 600 mg: Part I
Number analyzed (Participants) | 40 | 43 | 42 | 41 | 42
Percentage of participants | 85.0 [70.2 to 94.3] | 83.7 [69.3 to 93.2] | 92.9 [80.5 to 98.5] | 90.2 [76.9 to 97.3] | 81.0 [65.9 to 91.4]
Statistical Analysis 1: Comparison: Doravirine 25 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in % response = 4.5, 95% CI 2-sided [-12.5 to 21.5] — A positive value would be considered as favoring doravirine over efavirenz
Statistical Analysis 2: Comparison: Doravirine 50 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in % response = 2.8, 95% CI 2-sided [-13.9 to 19.8] — A positive value would be considered as favoring doravirine over efavirenz
Statistical Analysis 3: Comparison: Doravirine 100 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in % response = 12.2, 95% CI 2-sided [-2.5 to 28.0] — A positive value would be considered as favoring doravirine over efavirenz
Statistical Analysis 4: Comparison: Doravirine 200 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in % response = 9.5, 95% CI 2-sided [-6.2 to 25.7] — A positive value would be considered as favoring doravirine over efavirenz

11. Secondary Outcome: Percentage of Participants With Virologic Response (HIV-1 RNA <200 Copies/mL) at Week 24: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: Assessment of the virologic response to doravirine at 100 mg, compared to efavirenz, each in combination with TRUVADA, as measured by the percentage of participants with plasma HIV-1 RNA <200 copies/mL at Week 24. HIV RNA levels were determined using the Abbott RealTime HIV-1 Assay. The percentage of participants in any treatment group with a virologic response was primarily assessed for Weeks 0-24. The NC=F approach was used as the primary approach to handle missing data for this analysis of efficacy. This secondary outcome was analyzed for HIV-1 RNA <200 copies/mL in Part I & Part II combined.
Time Frame: Week 24
Population: The analyzed population consisted of all randomized participants who received at least one dose of blinded study treatment in either Part I or Part II, and had at least one post-randomization observation for the analysis of HIV-1 RNA (<200 copies/mL) at 24 weeks of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 107 | 108
Percentage of participants | 89.7 [82.3 to 94.8] | 87.0 [79.2 to 92.7]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference in % response = 2.7, 95% CI [-6.1 to 11.7] — A positive value would be considered as favoring doravirine over efavirenz

12. Secondary Outcome: Percentage of Participants With Virologic Response (HIV-1 RNA <200 Copies/mL) at Week 48: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: Evaluation of the antiretroviral activity of doravirine at 100 mg, compared to efavirenz, each in combination with TRUVADA for 24 weeks, as measured by the percentage of participants with HIV-1 RNA <200 copies/mL at Week 48. HIV RNA levels were determined using the Abbott RealTime HIV-1 Assay. This primary outcome was analyzed for RNA <200 copies/mL in Part I & Part II combined.
Time Frame: Week 48
Population: The analyzed population consisted of all randomized participants who received at least one dose of blinded study treatment in either Part I or Part II, and had at least one post-randomization observation for the analysis of HIV RNA (<200 copies/mL) at 48 weeks of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 108 | 107
Percentage of participants | 85.2 [77.1 to 91.3] | 85.0 [76.9 to 91.2]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference in % response = 0.1, 95% CI 2-sided [-9.7 to 9.9] — A positive value would be considered as favoring doravirine over efavirenz

13. Secondary Outcome: Percentage of Participants With Virologic Response (HIV-1 RNA <200 Copies/mL) at Week 96: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: Assessment of the virologic response to doravirine at 100 mg, compared to efavirenz, each in combination with TRUVADA, as measured by the percentage of participants with plasma HIV-1 RNA <200 copies/mL at Week 96. HIV RNA levels were determined using the Abbott RealTime HIV-1 Assay. The percentage of participants in any treatment group with a virologic response was primarily assessed for Weeks 0-96. The Non-Completer = Failure (NC=F) approach, in which participants who prematurely discontinued assigned treatment for any reason and were considered as failures thereafter, was used as the primary approach to handle missing data this analysis of efficacy. This primary outcome was analyzed for HIV-1 RNA <200 copies/mL in Part I & Part II combined.
Time Frame: Week 96
Population: The analyzed population consisted of all randomized participants who received at least one dose of blinded study treatment in either Part I or Part II, and had at least one post-randomization observation for the analysis of HIV-1 RNA (<200 copies/mL) at 96 weeks of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 108 | 108
Percentage of participants | 79.6 [70.8 to 86.8] | 75.9 [66.7 to 83.6]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference in % response = 3.9, 95% CI 2-sided [-7.3 to 15.0] — A positive value would be considered as favoring doravirine over efavirenz

14. Secondary Outcome: Change From Baseline in CD4 T Lymphocyte Cell Count at Week 24: Doravirine (All Doses) vs Efavirenz (Part I)
Description: Evaluation of the change from baseline in the CD4 cell count at Week 24 in participants receiving doravirine at all doses (25 mg, 50 mg, 100 mg, and 200 mg), compared with participants receiving efavirenz 600 mg. The Observed Failure (OF) approach was used to handle missing data, and the Baseline CD4 cell count was carried forward for participants who discontinued assigned treatment due to lack of efficacy.
Time Frame: Baseline, Week 24
Population: The analyzed population consisted of all randomized participants who received at least one dose of blinded study treatment in Part I, and had at least one post-randomization observation for the analysis of CD4 cell count at 24 weeks of study treatment.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Doravirine 25 mg: Part I | Doravirine 50 mg: Part I | Doravirine 100 mg: Part I | Doravirine 200 mg: Part I | Efavirenz 600 mg: Part I
Number analyzed (Participants) | 38 | 41 | 41 | 40 | 40
cells/mm^3 | 154.1 [115.1 to 193.1] | 112.9 [74.5 to 151.2] | 133.6 [100.4 to 166.8] | 140.7 [95.6 to 185.7] | 121.1 [73.3 to 169.0]
Statistical Analysis 1: Comparison: Doravirine 25 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in CD4 change = 33.0, 95% CI 2-sided [-28.1 to 94.0] — A positive value would be considered as favoring doravirine over efavirenz
Statistical Analysis 2: Comparison: Doravirine 50 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in CD4 change = -8.3, 95% CI 2-sided [-68.5 to 51.9] — A positive value would be considered as favoring doravirine over efavirenz
Statistical Analysis 3: Comparison: Doravirine 100 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in CD4 change = 12.5, 95% CI 2-sided [-44.6 to 69.5] — A positive value would be considered as favoring doravirine over efavirenz
Statistical Analysis 4: Comparison: Doravirine 200 mg: Part I vs Efavirenz 600 mg: Part I; Test type: Superiority or Other; Difference in CD4 change = 19.6, 95% CI 2-sided [-45.1 to 84.2] — A positive value would be considered as favoring doravirine over efavirenz

15. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 24: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: Assessment of the change from baseline in the CD4 cell count at Week 24 in participants receiving doravirine at 100 mg, compared with participants receiving efavirenz 600 mg. The OF approach was used to handle missing data, and the Baseline CD4 cell count was carried forward for participants who discontinued assigned treatment due to lack of efficacy.
Time Frame: Baseline, Week 24
Population: The analyzed population consisted of all randomized participants who received at least one dose of blinded study treatment in either Part I or Part II, and had at least one post-randomization observation for the analysis of CD4 cell count at 24 weeks of study treatment.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 106 | 101
cells/mm^3 | 152.3 [121.7 to 182.8] | 146.0 [113.1 to 178.8]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference in CD4 change = 6.3, 95% CI 2-sided [-38.2 to 50.8] — A positive value would be considered as favoring doravirine over efavirenz

16. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: Assessment of the change from baseline in the CD4 count at Week 48 in participants receiving doravirine at 100 mg, compared with participants receiving efavirenz 600 mg. The OF approach was used to handle missing data, and the Baseline CD4 cell count was carried forward for subjects who discontinued assigned treatment due to lack of efficacy.
Time Frame: Baseline, Week 48
Population: The analyzed population consisted of all randomized subjects who had baseline data, received at least 1 dose of blinded study medication in either Part I or Part II, and had at least 1 post-randomization observation for the analysis of CD4 cell count at 48 weeks of study treatment.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 102 | 100
cells/mm^3 | 191.9 [160.8 to 223.1] | 194.5 [163.2 to 225.9]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference in CD4 change = -2.6, 95% CI 2-sided [-46.5 to 41.3] — A positive value would be considered as favoring doravirine over efavirenz

17. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: A secondary endpoint in Part I/II combined was the change from baseline in the CD4 count at Week 96 in participants receiving doravirine at 100 mg, compared with participants receiving efavirenz 600 mg. The OF approach was used to handle missing data, and the Baseline CD4 cell count was carried forward for subjects who discontinued assigned treatment due to lack of efficacy.
Time Frame: Baseline, Week 96
Population: The analyzed population consisted of all randomized subjects who had baseline data, received at least 1 dose of blinded study medication in either Part I or Part II, and had at least 1 post-randomization observation for the analysis of CD4 cell count at 96 weeks of study treatment.
Measure: Mean (95% Confidence Interval); unit: cells/mm^3
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 95 | 93
cells/mm^3 | 259.2 [220.0 to 298.3] | 263.6 [218.1 to 309.1]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference in CD4 change = -4.4, 95% CI 2-sided [-64.0 to 55.1] — A positive value would be considered as favoring doravirine over efavirenz

18. Secondary Outcome: Percentage of Participants With At Least 1 AE in Weeks 0-48: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: A secondary outcome in Part I/II combined was the percentage of participants receiving doravirine at 100 mg, compared with participants receiving efavirenz 600 mg, who had at least 1 AE over 48 weeks of treatment. The percentage of participants in any treatment group with at least 1 AE was primarily assessed for Weeks 0-48.
Time Frame: Up to Week 48
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 108 | 108
Percentage of participants | 87.0 [79.2 to 92.7] | 89.8 [82.5 to 94.8]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference = -2.8, 95% CI 2-sided [-11.7 to 6.0] — A negative value would be considered as favoring doravirine over efavirenz

19. Secondary Outcome: Percentage of Participants With At Least 1 AE in Weeks 0-96: Doravirine 100 mg vs Efavirenz (Part I & Part II Combined)
Description: A secondary outcome in Part I/II combined was the percentage of participants receiving doravirine at 100 mg, compared with participants receiving efavirenz 600 mg, who had at least 1 AE over 96 weeks of treatment. The percentage of participants in any treatment group with at least 1 AE was primarily assessed for Weeks 0-96.
Time Frame: Up to Week 96
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Doravirine 100 mg: Part I/II (Combined) | Efavirenz 600 mg: Part I/II (Combined)
Number analyzed (Participants) | 108 | 108
Percentage of participants | 89.8 [82.5 to 94.8] | 96.3 [90.8 to 99.0]
Statistical Analysis 1: Comparison: Doravirine 100 mg: Part I/II (Combined) vs Efavirenz 600 mg: Part I/II (Combined); Test type: Superiority or Other; Difference = -6.5, 95% CI 2-sided [-14.1 to 0.3] — A negative value would be considered as favoring doravirine over efavirenz

ADVERSE EVENTS:
Time Frame: 96 weeks
Description: All Treated participants randomized to doravirine or efavirenz using an IVRS
Groups:
- Doravirine 25 mg (n=40): Doravirine 25 mg once daily plus TRUVADA once daily received in Part I
- Doravirine 50 mg (n=43): Doravirine 50 mg once daily plus TRUVADA once daily received in Part I
- Doravirine 100 mg (n=108): Doravirine 100 mg once daily plus TRUVADA once daily received in Part I & Part II (Combined)
- Doravirine 200 mg (n=41): Doravirine 200 mg once daily plus TRUVADA once daily received in Part I
- Efavirenz 600 mg: Part I (n=108): Efavirenz 600 mg once daily plus TRUVADA once daily received in Part I & Part II (Combined)
Arm/Group | Doravirine 25 mg (n=40) | Doravirine 50 mg (n=43) | Doravirine 100 mg (n=108) | Doravirine 200 mg (n=41) | Efavirenz 600 mg: Part I (n=108)
Serious Adverse Events (participants affected / at risk) | 4/40 | 1/43 | 11/108 | 3/41 | 13/108
Other Adverse Events (participants affected / at risk) | 31/40 | 35/43 | 78/108 | 36/41 | 82/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doravirine 25 mg (n=40) (N=40) | Doravirine 50 mg (n=43) (N=43) | Doravirine 100 mg (n=108) (N=108) | Doravirine 200 mg (n=41) (N=41) | Efavirenz 600 mg: Part I (n=108) (N=108)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Biliary dyskinesia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute hepatitis C (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cryptosporidiosis infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
B-cell unclassifiable lymphoma high grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Kaposi's sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peroneal nerve palsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bipolar I disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doravirine 25 mg (n=40) (N=40) | Doravirine 50 mg (n=43) (N=43) | Doravirine 100 mg (n=108) (N=108) | Doravirine 200 mg (n=41) (N=41) | Efavirenz 600 mg: Part I (n=108) (N=108)
Ear pain (Ear and labyrinth disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 5 (5) | 0 (0) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 1 (2) | 3 (3) | 4 (5) | 2 (2) | 5 (9)
Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 2 (2) | 0 (0) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 10 (10) | 4 (4) | 16 (18) | 5 (5) | 18 (20)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 6 (6)
Nausea (Gastrointestinal disorders) | 3 (3) | 7 (8) | 13 (16) | 9 (9) | 11 (12)
Vomiting (Gastrointestinal disorders) | 4 (4) | 1 (1) | 6 (7) | 1 (1) | 7 (8)
Fatigue (General disorders) | 7 (7) | 5 (7) | 6 (9) | 5 (7) | 7 (7)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 6 (7) | 0 (0) | 3 (4)
Acute sinusitis (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 1 (2)
Bronchitis (Infections and infestations) | 5 (7) | 3 (5) | 5 (5) | 5 (7) | 12 (13)
Conjunctivitis (Infections and infestations) | 1 (1) | 2 (2) | 6 (7) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 1 (2) | 2 (3) | 9 (10) | 2 (2) | 1 (1)
Influenza (Infections and infestations) | 6 (9) | 2 (2) | 3 (3) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (4) | 5 (12) | 19 (31) | 12 (17) | 13 (16)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 2 (3) | 3 (3) | 3 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 5 (5) | 5 (7) | 2 (2) | 3 (4)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 5 (7) | 3 (4) | 5 (7)
Syphilis (Infections and infestations) | 4 (6) | 1 (2) | 6 (7) | 6 (7) | 8 (9)
Tinea pedis (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 4 (4)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 2 (6) | 10 (14) | 3 (3) | 13 (19)
Accidental overdose (Injury, poisoning and procedural complications) | 4 (4) | 1 (3) | 4 (5) | 3 (10) | 5 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 6 (6) | 3 (3) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 5 (7) | 6 (7) | 2 (2) | 10 (14)
Anogenital warts (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 4 (5) | 2 (2) | 6 (6)
Dizziness (Nervous system disorders) | 5 (5) | 5 (6) | 16 (17) | 3 (3) | 32 (38)
Headache (Nervous system disorders) | 5 (6) | 6 (8) | 14 (27) | 7 (7) | 15 (26)
Somnolence (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 5 (6) | 9 (9) | 7 (9) | 4 (4) | 19 (21)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 3 (4) | 0 (0) | 6 (9)
Depression (Psychiatric disorders) | 1 (1) | 3 (4) | 4 (4) | 0 (0) | 11 (12)
Insomnia (Psychiatric disorders) | 1 (1) | 6 (6) | 10 (10) | 3 (4) | 6 (7)
Nightmare (Psychiatric disorders) | 1 (1) | 1 (1) | 9 (10) | 0 (0) | 10 (12)
Sleep disorder (Psychiatric disorders) | 1 (1) | 2 (2) | 6 (6) | 0 (0) | 8 (11)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (7) | 1 (1) | 3 (4) | 3 (3) | 6 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 3 (3)
Acne (Skin and subcutaneous tissue disorders) | 2 (2) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 4 (4) | 0 (0) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (6) | 6 (6) | 2 (2) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less